CLINICAL TRIAL: NCT06523907
Title: "Effectiveness of Basic Nursing Educational Interventions on Primary Healthcare Paramedics: A Quasi-Experimental Approach"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SINA Health Education and Welfare Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00005
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Education Training; Nursing Skills; Primary Healthcare; Education, Nursing
Keywords: Education status; nursing skills; Nurse; needle stick injury; safe injection administration
MeSH Terms: conditions — Needlestick Injuries | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control " Present Knowledge about the Basic Nursing skills" (No Intervention)
- Intervention " Educational Intervention from Registered Nurse" (Experimental)
  Interventions: Other: Intervention Basic Nursing skills; Other: Control Present Knowledge about basic nursing skill

INTERVENTIONS:
Other: Intervention Basic Nursing skills — Evaluating the effectiveness of the education program in improving paramedics' knowledge of essential nursing care principles, such as hygiene practice, infection control, safe administration of injection, blood draw, vital sign monitoring, respiratory rate
  Other Names: Educational Intervention
  Arms: Intervention " Educational Intervention from Registered Nurse"
Other: Control Present Knowledge about basic nursing skill — Assess the current and baseline knowledge status of the participants about the hygiene practice, infection control, safe administration of injection, blood draw, vital sign monitoring, respiratory rate
  Arms: Intervention " Educational Intervention from Registered Nurse"

SUMMARY:
Expected Significance of the Study:

Improved Patient Outcomes: Paramedics often serve as the first point of contact for patients in primary healthcare settings. Ensuring that they possess adequate knowledge and skills in basic nursing care can lead to improved patient outcomes, including better management of chronic conditions, reduced incidence of complications, and enhanced overall quality of care.

Enhanced Healthcare Delivery: By equipping paramedics with basic nursing care education, healthcare systems can optimize resource utilization and improve the efficiency of care delivery. Paramedics may be better equipped to handle a wider range of patient needs, reducing the burden on other healthcare professionals and streamlining the referral process.

Addressing Skills Gaps: Many paramedics receive training primarily focused on emergency medical care rather than comprehensive nursing skills. This research addresses an important gap in paramedic education by evaluating the effectiveness of additional training in basic nursing care, potentially filling a critical need in the healthcare workforce.

Professional Development: Providing paramedics with opportunities for ongoing education and professional development can enhance job satisfaction, increase retention rates, and contribute to a more skilled and competent workforce. This research could inform the development of training programs tailored to the specific needs of paramedics in primary healthcare settings.

Cost-Effectiveness: Investing in education and training programs for paramedics may yield long-term cost savings for healthcare systems by reducing hospital admissions, emergency department visits, and unnecessary medical interventions. Assessing the effectiveness of such programs is crucial for allocating resources effectively and maximizing their impact.

Evidence-Based Practice: By conducting a quasi-experimental study to evaluate the effectiveness of basic nursing care education among paramedics, this research contributes valuable evidence to the field of healthcare education and practice. Evidence-based findings can inform policy decisions, curriculum development, and clinical guidelines, ultimately benefiting both patients and healthcare providers.

DETAILED DESCRIPTION:
Nursing care is the cornerstone of primary healthcare organizations, playing a vital role in promoting health, preventing illness, and managing chronic conditions within communities. At the forefront of patient interaction, nurses in primary healthcare settings provide comprehensive and holistic care that addresses individuals' physical, emotional, and social needs. In these settings, nursing care encompasses a wide range of services, including health assessments, health education, disease prevention, and health promotion initiatives. Nurses collaborate closely with other healthcare professionals, such as physicians, pharmacists, and allied health workers, to deliver coordinated and patient-centered care.

Moreover, nursing care in primary healthcare organizations extends beyond individual patient encounters to encompass community-based initiatives and population health management strategies. Nurses engage in community outreach programs, health education workshops, and health promotion campaigns aimed at empowering individuals and communities to adopt healthy behaviors and lifestyles.

In essence, nursing care at primary healthcare organizations embodies the principles of accessibility, continuity, comprehensiveness, and patient-centeredness. Through their expertise, dedication, and advocacy, nurses contribute significantly to improving health outcomes and fostering wellness in the communities they serve.

Rationale:

Paramedics play a crucial role in primary healthcare, often being the first point of contact for patients in need of medical assistance. However, their training may not always encompass the depth of nursing care required in certain situations. This study seeks to bridge this gap by evaluating the outcomes of implementing a structured basic nursing care education program tailored to the needs of paramedics.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria include at least one year of working experience in the hospital, willingness to participate in the study, and not participating in similar training courses

Exclusion Criteria:

* The exclusion criteria include not attending more than two training sessions will exclude from the study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Pre and post assessment of Paramedics' Knowledge after educational intervention | One month
  Baseline knowledge about the primary healthcare settings among the paramedics before the intervention given

SECONDARY OUTCOMES:
Pre and Post Intramuscular injection administration Knowledge | One month
  Comparing the pre- and post-intervention knowledge among paramedics about how to administer I/V injection, who underwent the education program.
Pre and Post Intramuscular injection administration Knowledge | One month
  Identifying any barriers or challenges encountered in implementing the education program and suggesting recommendations for future improvements or modifications.
Pre and Post Sub-cutaneous injection administration knowledge | one month
  Investigating any changes in paramedics' attitudes towards nursing care, including their perceived importance of nursing interventions in primary healthcare contexts.
Pre and Post Needle Stick Injury administration Knowledge | one month
  Investigating any changes in paramedics' attitudes towards nursing care, including their perceived importance of nursing interventions in primary healthcare contexts.
Pre and Post educational intervention of Hygiene practice knowledge | one month
  Investigating any changes in paramedics' attitudes towards nursing care, including their perceived importance of nursing interventions in primary healthcare contexts.
Pre and Post educational intervention of vital sign knowledge | one month
  Investigating any changes in paramedics' attitudes towards nursing care, including their perceived importance of nursing interventions in primary healthcare contexts.
Pre and Post educational intervention of anthropometric measurement (weight in Kg) knowledge | one month
  Investigating any changes in paramedics' attitudes towards nursing care, including their perceived importance of nursing interventions in primary healthcare contexts.
Pre and Post educational intervention of anthropometric measurement (Height in cm) knowledge | one month
  Investigating any changes in paramedics' attitudes towards nursing care, including their perceived importance of nursing interventions in primary healthcare contexts.

CONTACTS AND LOCATIONS:
Locations (1):
- SINA Health Education & Welfare Trust, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared upon suitable request